CLINICAL TRIAL: NCT05704218
Title: Hypersensitivity Pneumonitis of Domestic Origin: Investigation of the Microorganisms Involved and Improvement of Serological Diagnosis.
Brief Title: Hypersensitivity Pneumonitis of Domestic Origin
Acronym: HOME-HP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/736
Record Dates: First submitted 2022-12-02; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2022-11

CONDITIONS: Sensitisation; Mold or Dust Allergy; Respiratory Disease
Keywords: hypersensitivity pneumonitis; molds; dwellings; thresholds
MeSH Terms: conditions — Respiration Disorders; Alveolitis, Extrinsic Allergic | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: the final diagnosis will be judged by the pneumologist on plural results: imagery, BALF cytology. The final diagnosis will be used to make 2 groups proven / non proven domestic forms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- domestic HP (Other): All the patients will be in the same arm until obtention of the final diagnosis.
  The final diagnosis will be used to compare data of serology to determine thresholds
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — the patient will have a blood sample in order to perform serology tests

SUMMARY:
Exposure to molds in dwellings is a public health problem. Diagnosis of hypersensitivity pneumonitis due to mold exposure at home (domestic HP) are increasing. To perform the serodiagnosis of domestic HP a cohort constitued of proven cases and exposed healthy controls are needed.

The HOME HP study aimed at obtaining a cohort of proven cases and exposed controls in order to be able to improve the serodiagnosis of domestic HP.

DETAILED DESCRIPTION:
Hypersensitivy pneumonitis (HP) are chronic respiratory diseases due to frequent exposure to high quantities of allergens (molds, bacteria, mycobacteria, avian proteins). In case of domestic HP, patients are exposed at home to molds due to flooding or poor ventilation.

The diagnosis of domestic HP includes detection of IgG towards molds. A prior study in 2005 allowed the determination of frequent allergenic molds isolated in homes in Bourgogne Franche Comte (study on 110 dwellings). However, no real cohort of proven cases versus controls is available. So, we are lacking validated thresholds. The HOME HP study is a prospective study that will include several centers of pneumology on France territory. The fungal contamination of dwellings occupied by patients suffering of interstitial disease (DIP), including suspicion of domestic HP, will be analyzed. The most frequently isolated molds will be then produced as antigens and will be tested in order to assess the sensitization of the included patients. The data of imagery, BALF cytology will allow to determine if patients are diagnosed with domestic HP or not. We will then obtain 2 groups of patients 1-proven domestic HP and 2-non domestic HP . Comparing the number of immunization arcs between the 2 groups will then be possible to validate appropriate thresholds for the serodiagnosis of domestic HP.

Domestic HP are rare diseases, so a high number of inclusions will be needed to obatin in 2 years about 25-30 proven cases. The HOME HP study is important to improve the serodiagnosis of domestic HP.

ELIGIBILITY:
Inclusion Criteria:

* exposure to mold at home
* given consent
* suspicion of doemstic HP
* clinical signs of interstial pneumopathy

Exclusion Criteria:

* immunocompromised patients
* prior diagnosis of another HP form (avian, farm, bath tub etc..)
* exposure to avian proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
measurement of mold sensitisation | 2 years
  serology
measurement of mold presence in dwellings | 2 years
  dust collectors
testing of new fungal antigens | 2 years
  ELISA

IPD SHARING:
Plan to Share IPD: No